CLINICAL TRIAL: NCT01258127
Title: Adjuvant Chemotherapy of Pemetrexed/Carboplatin Compared With Vinorelbine/Carboplatin in Patients With Completely Resected NSCLC
Brief Title: Pemetrexed/Carboplatin vs Vinorelbine/Carboplatin in Patients With Completely Resected Non-small Cell Lung Cancer (NSCLC)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shanghai Nancy Medical Sci-Tech Co. Ltd (Industry)
Collaborators: Sichuan Cancer Hospital and Research Institute (Other)
Responsible Party: Department of Thoracic Surgery, Cancer Hospital of Sichuan Province
Other Study IDs: PCVC001
Record Dates: First submitted 2010-12-09; First posted 2010-12-10 (Estimated); Last update posted 2010-12-10 (Estimated); Status verified 2010-12

CONDITIONS: Non-small Cell Lung Cancer
Keywords: Pemetrexed; Vinorelbine; Carboplatin
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Pemetrexed and Carboplatin: For patients in arm pemetrexed/carboplatin, folic acid (350-1000 μg) must be given daily beginning approximately 5-7 days prior to first dose of pemetrexed and continuing daily until 3 weeks after the last dose of study therapy. Vitamin B12 (1000 μg) will be administered as an intramuscular injection approximately 1 to 2 weeks prior to first dose of pemetrexed and repeated approximately every 9 weeks until 3 weeks after the last dose of study therapy. Dexamethasone (4 mg of oral or equivalent) given twice daily should be taken on the day before, the day of, and the day after each dose of pemetrexed, for rash prophylaxis unless medically contraindicated. Patients must receive pemetrexed at day 1 at the dose of 500 mg/m2 as an IV infusion over approximately 10 minutes, then carboplatin target area under the concentration curve (AUC) 6 (i.v. infusion over 30 minutes) on day 1 of a 21-day cycle. A total of four cycles is intended.
- Vinorelbine and Carboplatin: Patients in arm vinorelbine and carboplatin follow the regimen: The scheduled infusion time is 6-10 minutes for IV vinorelbine at the dose of 25 mg/m2 d1,8, then carboplatin target area under the concentration curve (AUC) 6 (i.v. infusion over 30 minutes) on day 1 of a 21-day cycle. A total of four cycles is intended.

SUMMARY:
The main purpose of this randomized phase II trial is to evaluate the clinical feasibility and activity of administering adjuvant chemotherapy of pemetrexed/carboplatin compared with vinorelbine/carboplatin in patients with completely resected non-small cell lung cancer (NSCLC).

DETAILED DESCRIPTION:
Pemetrexed, a multi-target folate antimetabolite, shows clear activity in non-small cell lung cancer (NSCLC). In a phase III study for patients with previously treated advanced NSCLC, the efficacy of single-agent pemetrexed, as determined by overall survival, was similar to that of docetaxel. (Hanna et al, 2004) The combination of carboplatin and pemetrexed has been of particular interest because it has demonstrated both good efficacy and a tolerable side effect profile. Phase I studies evaluated pemetrexed plus carboplatin in patients with malignant pleural mesothelioma, showed the regimen was efficacious and well tolerated. (Hughes et al, 2002) The combination of oxaliplatin and pemetrexed was compared with carboplatin and pemetrexed as first-line therapy for advanced NSCLC in a randomized phase II study. Response rates were 27 and 33%, respectively, and not statistically different. Toxicity in the carboplatin/pemetrexed arm was low, this doublet can be delivered easily and is well tolerated. Dose reductions occur only in 3.7% cycles. (Scagliotti et al, 2005) Therefore, it seems reasonable to test a less toxic regimen in patients with NSCLC after complete (R0) resection of the tumor, where reduced toxicities might improve the feasibility of drug delivery, compliance and the convenience of treatment for the patient and hence perhaps improve survival. The main purpose of this randomized phase II trial is to evaluate the clinical feasibility and activity of administering adjuvant chemotherapy of pemetrexed/carboplatin compared with vinorelbine/carboplatin in patients with completely resected NSCLC.

ELIGIBILITY:
Inclusion Criteria:

* Patients with completely resected stage IB (>4 cm), II, or IIIA non-squamous NSCLC. Patient must be enrolled and begin therapy within 4-6 weeks from the date of complete surgical resection.
* Fresh tissue must be available for genomics expression profiling.
* ECOG performance status of 0 or 1.
* No prior chemotherapy, radiation therapy, or biologic/targeted therapy within the last 5 years. Prior therapy with low dose methotrexate or similar medications is allowed if therapy used to treat non-malignant conditions.
* Age ≥18 years.
* No previous or concomitant malignancy in the past 5 years other than curatively-treated carcinoma in situ of the cervix, or basal cell or squamous cell carcinoma of the skin.
* No other serious medical or psychiatric illness.
* Signed informed consent.
* Required laboratory data within one week of enrollment: a)ANC or AGC ≥ 1500 per uL; b)Platelets ≥ 100,000 per uL; c)Total bilirubin ≤ 1.5 mg/dL; d)Creatinine < 2 mg/dL; creatinine clearance ≥ 45 mL/min; e)SGOT/SGPT ≤ 1.5× ULN.
* Females of child-bearing potential (not surgically sterilized and between menarche and 1 year post menopause) must test negative for pregnancy within 7 days prior to or at the time of enrollment based on a serum pregnancy test. Both sexually active males and females of reproductive potential must agree to use a reliable method of birth control, as determined by the patient and their health care team, during the study and for 3 months following the last dose of study drug.

Exclusion Criteria:

* Treatment within the last 30 days with a drug that has not received regulatory approval for any indication at the time of study entry.
* Concurrent administration of any other anti-tumor therapy.
* Inability to comply with protocol or study procedures.
* Active infection requiring IV antibiotics, antifungal or antiviral agents, that in the opinion of the investigator would compromise the patient's ability to tolerate therapy.
* Major surgery (other than definitive lung cancer surgery) within two weeks of study or other serious concomitant systemic disorders that, in the opinion of the investigator, would compromise the safety of the patient or compromise the patient's ability to complete the study.
* Myocardial infarction having occurred less than 6 months before inclusion, any known uncontrolled arrhythmia, symptomatic angina pectoris, active ischemia, or cardiac failure not controlled by medications.
* Contraindication to corticosteroids.
* Inability or unwillingness to take folic acid or vitamin B12 supplementation.
* Presence of clinically significant third-space fluid collections (for example, ascites or pleural effusions) that cannot be controlled by drainage or other procedures prior to study entry and throughout study enrollment as the distribution of pemetrexed in this fluid space is not fully understood.
* Inability to discontinue administration of aspirin at a dose > 1300 mg/day or other long acting, non-steroidal anti-inflammatory agents for 2 days before, the day of, and 2 days after the dose of pemetrexed (5 days prior for long-acting agents such as piroxicam). Moderate dose ibuprofen may be continued.
* Female patients that are pregnant or breast-feeding.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients are eligible to be included in the study only if they meet all of the following criteria.
Sampling Method: Probability Sample
Enrollment: 134 (Estimated)
Dates: Start 2010-08; Primary Completion 2012-08 (Estimated); Study Completion 2015-08 (Estimated)

PRIMARY OUTCOMES:
To determine the clinical feasibility rate (CFR) of 4 cycles of adjuvant chemotherapy with Pemetrexed and Carboplatin vs. Vinorelbine and Carboplatin | 1 month
  To determine the clinical feasibility rate (CFR) of 4 cycles of adjuvant chemotherapy with Pemetrexed and Carboplatin vs. Vinorelbine and Carboplatin in patients with NSCLC stage IB, IIA, IIB and T3N1 (without need for further radiotherapy). Treatment is considered to have clinical feasibility if dose limiting toxicity (DLT) will not be observed, and no non-acceptance by the patient leading to premature withdrawal, and no death due to cancer or cancer therapy will occur.

SECONDARY OUTCOMES:
To determine and compare the drug delivery between both treatment arms | 1 month
The relapse free survival | 3 months
The overall survival | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Hospital of Sichuan Province, Chengdu, Sichuan, China